CLINICAL TRIAL: NCT00870844
Title: A Randomised, Double-blind, Placebo-controlled, Multiple-dose, Dose-escalation Study of the Safety, Tolerability, and Pharmacokinetics of Lu AA24493 in Patients With Acute Ischemic Stroke
Brief Title: Safety and Pharmacokinetic Study of Carbamylated Erythropoietin (CEPO) to Treat Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12053A; 2007-003390-81 (EudraCT Number)
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Erythropoietin; Carbamylated; Neuroprotection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lu AA24493 (CEPO): 0.5 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Lu AA24493 (CEPO): 5.0 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Lu AA24493 (CEPO): 50.0 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AA24493 (CEPO) — 0.5 to 50.0 mcg/kg body weight, IV, within 0 to 48 hrs from symptom onset
  Arms: Lu AA24493 (CEPO): 0.5 mcg/kg; Lu AA24493 (CEPO): 5.0 mcg/kg; Lu AA24493 (CEPO): 50.0 mcg/kg
Drug: Placebo — Vials with solution for IV infusion
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to determine whether carbamylated erythropoietin (CEPO) dosed once daily for 5 days is a safe treatment for patients who have suffered an acute ischemic stroke.

DETAILED DESCRIPTION:
Acute ischemic stroke is a major cause of death and severe disability. The naturally occurring hormone, erythropoietin (EPO), is able to protect various neuronal tissues from ischemic injury and is beneficial in animal models of acute ischemic stroke. Lu AA24493 is a modified (carbamylated) version of EPO, neuroprotective but without the haematopoietic side effects. Lu AA24493 is developed for treatment of patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 90 years
* Clinical diagnosis of acute ischemic stroke
* Measurable stroke-related deficit
* Patient is stable
* Treatment can be initiated between 0 hours and 48 hours after the onset of stroke
* Expected hospital stay of at least 120 hours after first dose of study medication
* If female then not of childbearing potential

Exclusion Criteria:

* Primary intracerebral haemorrhage (ICH), or parenchymal haemorrhagic transformation of infarction (type PHI or PHII as defined in ECASS), subarachnoid haemorrhage (SAH), arterio-venous malformation (AVM), cerebral aneurysm, or cerebral neoplasm
* Treated with a thrombolytic <24 hours (if >24 hours and excluded ICH then eligible)
* Score >=1 on the NIHSS item 1a
* Pre-stroke mRS score >=2
* Uncontrolled hypertension
* Previous treatment with erythropoietin
* Previous exposure to Lu AA24493

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) and the modified Rankin Scale (mRS) | NIHSS = Baseline: Day 2, 3, 4, 5, Day 6/Discharge, Day 14, 30. mRS = Baseline, Day 6/Discharge, Day 14, 30

SECONDARY OUTCOMES:
Pharmacokinetics, immunogenicity and biomarkers | Baseline, Days 1-6, Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (5):
- FI004, Helsinki, Finland
- FR002, Paris, France
- NL005, Breda, Netherlands
- SG003, Singapore, Singapore
- GB001, Glasgow, United Kingdom